CLINICAL TRIAL: NCT03399981
Title: An Observational Study Utilising Data From the US Tysabri TOUCH Programme and Select EU MS Registries to Estimate the Risk of Progressive Multifocal Leukoencephalopathy (PML) and Other Serious Opportunistic Infections Among Patients Who Were Exposed to an MS Disease Modifying Treatment Prior to Treatment With Tysabri
Brief Title: Tysabri Observational Cohort Study - Multiple Sclerosis (MS) Registries
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 101MS411; EUPAS19800 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Progressive Multifocal Leukoencephalopathy
MeSH Terms: conditions — Leukoencephalopathy, Progressive Multifocal | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tysabri (TOUCH Cohort): Participants from the Tysabri TOUCH prescribing programme who have switched to Tysabri from newer DMTs (including fingolimod, dimethyl fumarate and teriflunomide) and the established DMTs (interferon beta and glatiramer acetate).
  Interventions: Biological: Tysabri
- Tysabri (EU MS Cohort): Participants from the EU MS registry who have switched to Tysabri from newer DMTs (including fingolimod, dimethyl fumarate and teriflunomide) and the established DMTs (interferon beta and glatiramer acetate).
  Interventions: Biological: Tysabri

INTERVENTIONS:
Biological: Tysabri — Administered as specified in the treatment arm.
  Other Names: Natalizumab BG00002

SUMMARY:
The primary purpose of this study is to estimate the incidence of progressive multifocal leukoencephalopathy (PML) among patients who switched to Tysabri from disease modifying therapies (DMTs), including newer DMTs (including fingolimod, dimethyl fumarate and teriflunomide) and the established DMTs (interferon beta and glatiramer acetate). Researchers will also look to estimate the incidence of other serious opportunistic infections among patients who switch to Tysabri from newer DMTs (including fingolimod, dimethyl fumarate and teriflunomide) and the established DMTs (interferon beta and glatiramer acetate)

DETAILED DESCRIPTION:
This is an observational cohort study utilising all available data from the Tysabri TOUCH (TYSABRI Outreach: Unified Commitment to Health) prescribing programme (US) supplemented with data from European Union (EU) multiple sclerosis (MS) registries to estimate the risk of PML and other serious opportunistic infections (OIs) among patients on Tysabri who have switched from newer DMTs (including fingolimod, dimethyl fumarate and teriflunomide) and the established DMTs (interferon beta and glatiramer acetate).

This study will provide cumulative data from its two components: a retrospective component (data captured prior to 01 January 2016) and a prospective component (data captured, and patients followed up, from 01 January 2016 through 31 December 2023; total prospective study duration of 8 years). All patients who switched to Tysabri from another DMT through 31 December 2020 will be included. The study will continue to follow-up patients until 31 December 2023 to allow for a minimal follow-up of 3 years.

ELIGIBILITY:
Key Inclusion Criteria:

* All TOUCH and available EU MS registry participants who have switched from DMTs (including fingolimod, dimethyl fumarate, teriflunomide, interferon beta and glatiramer acetate) and have one or more infusion(s) of Tysabri.

Key Exclusion Criteria:

* Not applicable

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All TOUCH and available EU MS registry participants who have switched from DMTs (including fingolimod, dimethyl fumarate, teriflunomide, interferon beta and glatiramer acetate) and have one or more infusion(s) of Tysabri.
Sampling Method: Non-Probability Sample
Enrollment: 80327 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Prospective and Retrospective Analyses: Number of Participants with Confirmed Progressive Multifocal Leukoencephalopathy (PML) | Retrospective: from the time of switching to Tysabri to 31 December 2015; Prospective: from the time of switching to Tysabri (on or after 01 January 2016) to 31 December 2023 (up to 8 years)
  Confirmed cases of PML must have one of the following:
  • Brain biopsy or brain from post mortem examination showing evidence of viral cytopathic changes on hematoxylin and eosin (H & E) staining associated with either positive immunohistochemistry for SV40 or in-situ hybridization for John Cunningham Virus (JCV) deoxyribonucleic acid (DNA) OR
  All of the following criteria:
  • Cerebrospinal fluid (CSF) with evidence of JCV DNA, preferably by ultra-sensitive quantitative polymerase chain reaction (PCR) testing (limit of quantification of ≤ 50 copies/ml), or JCV DNA on brain biopsy by PCR AND detailed description of brain magnetic resonance imaging (MRI) findings that are consistent with PML AND PREFERABLY new or progressive clinical symptoms suggestive of PML
Prospective and Retrospective Analyses: Number of Participants with Serious Adverse Events of Other Serious Opportunistic Infections (OIs) | Retrospective: from the time of switching to Tysabri to 31 December 2015; Prospective: from the time of switching to Tysabri (on or after 01 January 2016) to 31 December 2023 (up to 8 years)
  An SAE is any untoward medical occurrence at any dose that results in death, immediate risk of death, hospitalization, disability, or congenital anomaly/birth defect.
  Opportunistic infections (OIs) are infections that occur more frequently and are more severe in individuals with weakened immune systems.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Cambridge, Massachusetts, United States